CLINICAL TRIAL: NCT03540966
Title: Development and Psychometric Validation of the Chinese Version of Vitiligo Life Quality Index and Effects of Camouflage on the Life Quality of Patients With Vitiligo: A Randomized Open-label Controlled Study
Brief Title: Effects of Camouflage on the Life Quality of Patients With Vitiligo
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: XJPF-LCY-V201804
Record Dates: First submitted 2018-05-04; First posted 2018-05-30 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-03

CONDITIONS: Quality of Life

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): complete Chinese version of the vitiligo life quality index, VLQI-C, conventional therapies plus CapulinTM on-demand treatment period
  Interventions: Combination Product: CapulinTM; Other: Chinese version of the vitiligo life quality index, VLQI-C
- Group B (Placebo Comparator): complete Chinese version of the vitiligo life quality index, VLQI-C, conventional therapies on-demand treatment period
  Interventions: Other: Chinese version of the vitiligo life quality index, VLQI-C

INTERVENTIONS:
Combination Product: CapulinTM — a kind of camouflage agent
  Arms: Group A
Other: Chinese version of the vitiligo life quality index, VLQI-C — a questionaire designed for patients with vitiligo

SUMMARY:
Vitiligo is a common depigmented skin disease characterized by destruction of functional melanocyte.The recent therapies to vitiligo are including oral or external glucocorticoids, antioxidants, calcineurin inhibitors or phototherapy. However, long treatment period and unsatisfactory curative effects still exist, which confer long-term psychological burden to patients. As above concerns, it is of great value to explore therapeutic methods that can effectively control disease, improve appearance, relieve patients' pain and improve their quality of life. Current problem is the lack of a vitiligo life quality evaluation scale with Chinese characteristics for us. Therefore, it is necessary for the investigator to compile a vitiligo quality of life scale that is simple, feasible and applicable to China's national conditions. Meanwhile the reliability analysis must be carried out to bring better quality of life assessment tools to patients with vitiligo in China. Previous studies recommended that CapulinTM showing a good cover effect on vitiligo, but the effects of camouflage on the QoL of patients with vitiligo in Chinese population is unknown. Thus, the investigators undergo a randomized open-label controlled study to estimate the effects of CapulinTM on QoL of patients with vitiligo.

DETAILED DESCRIPTION:
Vitiligo is a common depigmented skin disease characterized by destruction of functional melanocyte. The global incidence is about 0.5-2.0% and prevalence be about 0.8-1.5% in China. Studies showed that almost half of vitiligo patients had developed depigmentation before 20 years old. Lesions involving exposed skin such as face, hand or mucous always make patients feeling embarrassment, so the impaired quality of life (QoL) have greater impact on patients with vitiligo than the disease itself. Besides, Vitiligo is also a psychosomatic disease as its cause stress or depression which can induce dysfunction of endocrine system or immune system in patients, finally resulted in poor curative effects and relapse of the disease which further aggravates stress and depression in patients. Furthermore, traditional Chinese medicine suggested that uneasiness would be a cause of vitiligo as well.

It is of great value to explore therapeutic methods that can effectively control disease, improve appearance, relieve patients' pain and improve their quality of life. Dermatologists of Japan and European suggested that camouflage would be a proper way to improve patients' appearance and it should be an effective supplement to the treatments of vitiligo.

With the transformation of the medical model from a simple biomedical model to a bio-psychological-social medical model, observing changes of lesion in vitiligo may not fully reflect the impact of vitiligo on patients. Therefore, it is necessary to develop some evaluation methods to reflect the impact of vitiligo in patients. Among the various measurement tools, universality scales have a wide range of measurement and can be applied to different groups of people to understand the general health status of the general population. But there are some limitations due to the unspecifically designed for a disease group. When the universal scale is applied to a specific disease, it does not have specificity. Some clinically significant information on quality of life may be omitted, and the QOL cannot be sensitively reflected. The scales in the dermatology area were developed for patients with dermatological diseases and reflect the differences between skin diseases and other system diseases. However, the specificity and sensitivity of specific diseases are still not strong enough.The problem is the lack of a vitiligo life quality evaluation scale with Chinese characteristics for us. Therefore, it is necessary for the investigator to compile a vitiligo quality of life scale that is simple, feasible and applicable to China's national conditions. Meanwhile the reliability analysis must be carried out to bring better quality of life assessment tools to patients with vitiligo in China.

Camouflage is an emerging solution to improve patients' appearance which showing a great potential in treatment of vitiligo. Diagnosis and treatment of vitiligo consensus (2014 edition) made by the dermatological department of the Chinese medical association also suggest that camouflage can be used on exposed skin such as face, neck, hands or feet.The first commercial camouflage agent in China is CapulinTM by 2004, Its formula contains natural plant extracts, moisturizers, emollients and natural pigments. The regimented mechanism is to combine the camouflage with the free protein on the cuticle and finally format the mimic human natural melanin, which is extremely similar to normal skin tone. Previous studies recommended that CapulinTM showing a good cover effect on vitiligo, but the effects of camouflage on the QoL of patients with vitiligo in Chinese population is unknown. Thus, the investigators undergo a randomized open-label controlled study to estimate the effects of CapulinTM on QoL of patients with vitiligo.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who signed Informed Consent Form；
* Male or female subjects 18-64 years of age；
* Clinically confirmed diagnosis of vitiligo as per the diagnostic criteria for vitiligo specified in Clinical Dermatology.

Exclusion Criteria:

* Incompliance with the diagnosis of vitiligo.
* Patients who had used other camouflage before;
* Cannot read or understand questionnaire.
* Patients who had taken antidepressants in the last three months had psychiatric and psycho-related illnesses.；
* Inability to guarantee taking medications and completing visits as scheduled during the study;
* Allergic history of any relevant ingredient in the camouflage;
* The combination of eczema, contact dermatitis, urticaria and other allergic diseases or other serious diseases which are not suitable for the treatment of skin diseases；
* Serious life-threatening condition such as cancer, autoimmune diseases；
* Women of child-bearing potential who are pregnant, plan to become pregnant during study or are lactating；
* Participating in other clinical studies or within 3 months;
* Any other condition that the investigator deems unsuitable for entering the study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Chinese version of the vitiligo life quality index, VLQI-C | 4 weeks
  Chinese version of the vitiligo life quality index, VLQI-C

SECONDARY OUTCOMES:
VASI Scoring Criteria | 4 weeks
  VASI=Σall body sites (hand units) × depigmentation
Vitiligo European Task Force assessment, VETFa | 4 weeks
  Vitiligo European Task Force assessment, VETFa

CONTACTS AND LOCATIONS:
Overall Officials: Chunying Li, Principal Investigator — Principal Investigator
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chang Y, Zhang S, Zhang W, Li S, Li C. The Efficacy and Psychoneuroimmunology Mechanism of Camouflage Combined With Psychotherapy in Vitiligo Treatment. Front Med (Lausanne). 2022 May 27;9:818543. doi: 10.3389/fmed.2022.818543. eCollection 2022. PMID 35721084